CLINICAL TRIAL: NCT01735435
Title: Tight Caloric Balance in Geriatric Patients After Hip Fracture.
Brief Title: Tight Caloric Balance in Geriatric Patients
Acronym: TICACOSiGP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Pierre singer, Professor Pierre Singer, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5744
Record Dates: First submitted 2012-11-24; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Nutrition Assessment
Keywords: geriatric patients; nutritional support
MeSH Terms: interventions — Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Control group) (No Intervention): Group 2(Control group)-patients in this group received nutrition according to the standard hospital dietary regimen.
- Group 1 (Indirect Calorimetry) (Experimental): Group 1(Indirect Calorimetry)-The tight calorie group received calories with an energy goal determined by repeated REE measurements using indirect calorimetry.
  Interventions: Other: Indirect Calorimetry

INTERVENTIONS:
Other: Indirect Calorimetry — The tight calorie group received calories with an energy goal determined by repeated REE measurements using indirect calorimetry.
  IC measurements:after a fasting period of at least 6 hours at three time periods : on admission to the study,between 24-48 hours following surgery and on the 7th day of the study.Measurements were performed by an experienced nurse or dietician,the device was automatically calibrated before each measurement and the REE was recorded after 15 minutes.
  Other Names: Energy intake according to REE measurements(nutrition according to the individual energy requirements)
  Arms: Group 1 (Indirect Calorimetry)

SUMMARY:
The aim of this study to assess the impact of nutritional support guided by repeated measurements of REE in geriatric patients following surgery for hip fractures.

Our hypothesis is that tight caloric control will reduce the risk of significant postoperative complications in geriatric patients following surgery for hip fractures.

Study Design :Prospective, Single center, Randomized, Unblinded study. Study Population:geriatric patients following surgery for hip fractures.

DETAILED DESCRIPTION:
The primary outcome:

presence of postoperative complications,hospital length of stay.

Secondary outcomes:

energy intake and calculated energy balance

Study Procedure:

eligible patients will be randomly assigned to 2 groups: the tight calorie (intervention)group and the control group.

ELIGIBILITY:
Inclusion Criteria:

patients older than 65 years who were admitted to the unit following hip fracture within 48 hours of the injury and in whom orthopedic surgery was considered the treatment of choice.

Exclusion Criteria:

Patients were excluded if they presented to hospital > 48 hours after the injury, were receiving steroids and/or immunosuppression therapy; in the presence of active oncologic disease, multiple fractures, diagnosed dementia or in the event that patients required supplemental nasal oxygen which precludes the measurement of resting energy expenditure.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Rate of postoperative complications | up to day 14
  incidence of postoperative complications following admission up to day 14/or hospital discharge and length of hospital stay will be evaluated

SECONDARY OUTCOMES:
Energy balance | prior to surgery and up to 14 day
  energy intake and calculated energy balance.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, Professor,MD, Principal Investigator — RabinMC,Beilinson Hospital
Locations (1):
- RabinMC, Petah Tikva, Israel